CLINICAL TRIAL: NCT04343924
Title: Clinical Study: Physiological Effects of Scuba Diving on PTSD by Activating the Parasympathetic System and Restoring the Optimal and Sustainable State of Balance Between the Sympathetic and Parasympathetic Autonomous Nervous System (Sympatho-vagale Scale)
Brief Title: Clinical Study About the Effects of Scuba Diving on Post Traumatic Stress Disorder (PTSD)
Acronym: DIVE4NICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-PP-12
Record Dates: First submitted 2020-04-03; First posted 2020-04-14 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Post-traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Diving Group (Experimental): The subjects of this group daily dive, 5 days per week, for a total of 10 dives at a maximum depth of 6 meters for a maximum duration of 20 minutes in a swimming pool.
  Interventions: Other: Scuba diving activities
- Virtual reality Group (Active Comparator): The subjects of this group will follow virtual reality sessions recreating the environment in which the submarine diver of the GP+ group operates.
  Interventions: Other: Virtual reality activities
- Control Group (No Intervention): The subjects of this group will be monitored and treated for PTSD and will not attend the dive discovery course or virtual reality sessions.

INTERVENTIONS:
Other: Scuba diving activities — The subjects of this group daily dive, 5 days per week, for a total of 10 dives at a maximum depth of 6 meters for a maximum duration of 20 minutes in a swimming pool.
  Arms: Diving Group
Other: Virtual reality activities — The subjects of this group will follow virtual reality sessions recreating the environment in which the submarine diver of the GP+ group operates
  Arms: Virtual reality Group

SUMMARY:
Post-traumatic stress disorder (PTSD) is a set of symptoms that can be developed as a result of exposure to a traumatic event or events that can range in prevalence from 25% to 75%. While therapeutic management combines psychotherapy, drug therapy and social support, some PTSD remain resistant after early and appropriate initial treatment. In terms of physiopathology, several studies have shown that parasympathetic activity is significantly decreased in patients with PTSD. In scuba diving, the cardio-vascular stresses associated with submersion of the subject and the lungs due to breathing in a regulator are at the origin of a reflex activation of the parasympathetic nervous system. The objective is to study the effects of the scuba diving activities-induced autonomic parasympathetic nervous system activation on the symptomatic progression of patients with PTSD.

The study population will consist of patients monitored and treated for PTSD following the attacks of 14/07/2016 in Nice (France).

DETAILED DESCRIPTION:
A group will be composed of patients (n=12) who will complete a Scuba Diving Discovery Course (GP+ Diving Group). This course, lasting 2 weeks, will consist of a daily dive, 5 days per week, for a total of 10 dives. These will be supervised by a graduate instructor according to the rules of supervision defined by the sport code. The dives will be conducted in open air, at a maximum depth of 6 meters for a maximum duration of 20 minutes.

A matched group (gender, age, height, weight and BMI) will be composed of patients (n=12) who will not complete the Scuba Diving Discovery Course (GP- Virtual reality group). The subjects of this group will follow virtual reality sessions recreating the environment in which the scuba divers of the GP+ group operate. A control group (GT) will be composed of patients (n=12) who are monitored and treated for PTSD and who will not attend the dive discovery course or virtual reality sessions.

* The main evaluation criterion will be the NON-INVASIVE determination of salivary alpha amylase.
* Secondary evaluation criteria will be heart rate variation, CGI, HAD and BECK Anxiety, EGF, PCL-S and IES questionary.

The main objective is to study the effects of immersion and pressure relief ventilation on the activation of the autonomic parasympathetic nervous system.

Secondary objectives are to assess the symptomatic impact of parasympathetic autonomic nervous system activation on overall improvement, anxiety and depressive symptoms, functioning, and the 3 subtypes of PTSD symptoms as vegetative neuro hyperactivity, invasive syndrome and avoiding

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Patients who understand and read French
* Patients who have signed the informed consent form
* Patients who have never practiced scuba diving
* Patients medically fit for scuba diving
* Patients with the DSM-5 criteria for Post-traumatic Stress Disorder
* PCL-S score strictly greater than 44
* CGI greater than or equal to 4
* Chronicity (duration greater than 3 months)

Exclusion Criteria:

* Women of reproductive age without contraception
* Pregnant or nursing women
* Patients under guardianship or curatorship and detainees of justice
* Patients who previously practised scuba diving or hold a diving certificate
* Patients whose medical condition medically contraindicated the practice of scuba diving,
* Patients having a water phobia, bipolar or psychotic disorder
* Patients with a severe and proven suicidal risk (MINI-S and medical examination)
* Patients treated for less than 2 months with antidepressants;
* Patients treated for less than 2 months with specific psychotherapy (Cognitive and Behavioural Therapy, EMDR)
* Patients with response to treatment (50% decrease in symptoms)
* Contraindications to the practice of virtual reality.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
The main objective is to study the physiological effects of pressure regulator immersion | 6 months
  Measure of parterial pressure
The main objective is to study the physiological effects of regulator ventilation on the activation of the parasympathetic autonomic nervous system | 6 months
  Measure of O2 saturation

CONTACTS AND LOCATIONS:
Overall Officials: Carl WILLEM, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No